CLINICAL TRIAL: NCT02353143
Title: First in Man Study With MEN1112, a CD157 Targeted Monoclonal Antibody, in Relapsed or Refractory Acute Myeloid Leukemia.
Brief Title: Study of MEN1112 Intravenous Infusion in Relapsed or Refractory Acute Myeloid Leukemia
Acronym: ARMY
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor accepted the iDSMB recommendation to terminate the study due to evidence of unpredictable liver toxicity and meaningful target engagement not translating into any clinical objective response.
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARMY-1; 2014-002433-59 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-02-02 (Estimated); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse
Keywords: Acute Myeloid Leukemia; AML; Relapsed; Refractory; MEN1112; Monoclonal antibody
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Intervention Model Description: The study included ascending doses in the range 0.1 mg/kg to 2.5 mg/kg. According to the Data Safety Review Board, doses to be sequentially tested are 0.1, 0.3, 0.6, 1, 1.7, 2.5 mg/kg single shot and 1.7, 2, and 3 mg/kg ramp up
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEN1112 (Experimental): Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation
  Interventions: Drug: MEN1112

INTERVENTIONS:
Drug: MEN1112 — Intravenous infusion of MEN1112 pro/Kg body weight dose will be administered for two 21-day cycles; MEN1112 dose is administered as' one shot infusion' (first group of patients) and as a dose to be infused in 3 days for the first two doses in Cycle 1 (second group of patients).
  Two treatment cycles will be followed by a 4-week End of Treatment Period and a Follow-up period. The individual treatment/observation period is six months (except for female patients of childbearing potential that will undergo monthly pregnancy test until 6 months from the last study drug administration).

SUMMARY:
The purpose of this study is to assess the safety of MEN1112, given as intravenous infusion, in patients with relapsed or refractory AML. Pharmacokinetics, clinical activity and potential immunogenicity of MEN1112 will be evaluated as well.

DETAILED DESCRIPTION:
This trial is designed as an open label, non randomised, dose escalation and cohort expansion, first administration to human study to be conducted in approximately 20 European sites. The study is aiming to identify the Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD), to assess the pharmacokinetics and to determine the clinical activity and potential immunogenicity of MEN1112, administered as IV infusion for two 21-day cycles.

Approximately 100 male and female ≥ 18 years-old patients, with a documented diagnosis of relapsed or refractory AML (not M3 FAB subtype), will be treated in the study, which consists of two steps.

Step 1 is the dose escalation phase according to a 3+3 patients cohort design. Incremental mg/Kg doses will be tested. Briefly, MEN1112 doses are to be administered to 3 patients; if no DLT is observed in a cohort of 3 DLT evaluable patients at a given dose level, the next cohort of 3 new patients will be treated with the next higher dose. In case of DLT occurrence by one of the three patients at any dose, the cohort will be expanded to 6 DLT evaluable patients at the same dose level. If two or more patients at a given dose level exhibit DLT, the dose escalation phase will be concluded as the MTD will be identified as one dose level below the one at which ≥ 2 DLT out of 6 treated patients occur.

Step 2 is the cohort expansion phase which will include patients treated at the MTD or the maximum dose level judged to be tolerable.

In each study Step, patients will be given two induction cycles of MEN1112 followed by a four-week End of Treatment period and a Follow-up period. In Step 1 and Step 2, DLT and MTD will be assessed when MEN1112 is given as a 'one shot' infusion (first group of patients) for all doses as well as a 'ramp up' administration to be infused in 3 days for the first two doses in Cycle 1 (second group of patients).

Along the study period, adverse events, changes in hematology/serum biochemistry parameters and bone marrow treatment response will represent the major clinical findings to be monitored on regular basis. The individual experimental clinical phase will last up to 6 months (except for female patients of childbearing potential that will undergo monthly pregnancy test until 6 months from the last study drug administration) encompassing approx. 40 planned visits at site, including Screening,Treatment, End of Treatment, Follow-up period and the End of Study visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years.
* Documented definitive diagnosis of AML (according to WHO criteria, 2008) that is relapsed/refractory to standard treatment, for which no standard therapy is available or the patient refuses standard therapy.
* WBC count ≤ 10 x 109/L at Visit 1/Day 1; hydroxyurea is allowed to lower WBC count.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at Visit1/Day 1.
* Life expectancy of at least 2 months.
* Adequate renal and hepatic laboratory assessments: Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered due to leukemic organ involvement, Total Bilirubin ≤2.0 × ULN, Serum creatinine ≤2.0 × ULN.
* Able to give written informed consent before any study related procedure

Exclusion Criteria:

* Acute promyelocytic leukaemia (French-American-British M3 classification).
* Active central nervous system involvement.
* Haematopoietic stem cell transplantation (HSCT) performed within 3 months prior to Screening Visit.
* Active infection requiring intravenous antibiotics.
* Life-threatening illnesses other than AML, uncontrolled medical conditions or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety or interfere with the patient's ability to comply with the study activities.
* Anti-tumour therapy within 14 days of study Visit 1/Day 1, excluding hydroxyurea.
* Prior participation in an investigational study (procedure or device) within 21 days of study Visit 1/Day 1.
* Radiotherapy within 28 days prior to study Visit 1/Day 1 or scheduled along the study conduct.
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Other active malignancies. History of malignancy in the last 12 months (except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast or non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Venditti, Professor, MD, Study Chair — Hematology Department, "Tor Vergata" University Viale Oxford, 81 00133 Rome, Italy
Locations (29):
- Belgium (5):
  - Antwerp
  - Brussels
  - Liège
  - Roeselare
  - Yvoir
- France (9):
  - Grenoble
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Paris
  - Pierre-Bénite
  - Toulouse
  - Villejuif
- Germany (4):
  - Dresden
  - Essen
  - Frankfurt
  - Munich
- Italy (5):
  - Bologna
  - Brescia
  - Milan
  - Rome
  - Torino
- Spain (6):
  - Badalona
  - Barcelona
  - Pamplona
  - Salamanca
  - Seville
  - Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: MEN1112 given as "one shot" infusion at the dosage of 0.1 mg/kg
- Cohort 2: MEN1112 given as "one shot" infusion at the dosage of 0.3 mg/kg
- Cohort 2b: MEN1112 given as "one shot" infusion at the dosage of 0.6 mg/kg
- Cohort 3: MEN1112 given as "one shot" infusion at the dosage of 1.0 mg/kg
- Cohort 3b: MEN1112 given as "one shot" infusion at the dosage of 1.7 mg/kg
- Cohort 3c: MEN1112 given as "one shot" infusion at the dosage of 2.5 mg/kg
- Cohort 1.7: MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg
- Cohort 2.0: MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg
- Cohort 3.0: MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Started (number of patients treated) | 4 | 7 | 6 | 8 | 26 | 5 | 3 | 8 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 7 | 6 | 8 | 26 | 5 | 3 | 8 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 2 | 1 | 2 | 4 | 13 | 2 | 2 | 2 | 1
Not completed — reason not specified | 1 | 2 | 0 | 0 | 6 | 1 | 0 | 3 | 1
Not completed — Physician Decision | 0 | 4 | 2 | 3 | 4 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — patient receiving other treatment for AML | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Dose limiting toxicity (DLT) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0 | Total
Number analyzed (Participants) | 4 | 7 | 6 | 8 | 26 | 5 | 3 | 8 | 4 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 5 | 3 | 7 | 0 | 3 | 6 | 2 | 32
  >=65 years | 3 | 2 | 1 | 5 | 19 | 5 | 0 | 2 | 2 | 39
Age, Continuous [Mean (Full Range); unit: years] | 69 [64 to 78] | 55.6 [20 to 76] | 53.8 [33 to 72] | 68.6 [56 to 77] | 69.2 [47 to 85] | 77.6 [71 to 87] | 58.3 [54 to 63] | 49.1 [19 to 71] | 56.8 [35 to 79] | 63.6 [19 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 4 | 12 | 4 | 1 | 4 | 2 | 32
  Male | 3 | 5 | 4 | 4 | 14 | 1 | 2 | 4 | 2 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 8
  Not Hispanic or Latino | 4 | 7 | 6 | 8 | 17 | 5 | 3 | 8 | 4 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 0 | 2 | 1 | 6 | 0 | 2 | 2 | 1 | 18
  Italy | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
  France | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3 | 6
  Germany | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 2 | 0 | 8
  Spain | 0 | 5 | 4 | 4 | 18 | 0 | 1 | 4 | 0 | 36
Weight [Mean (Full Range); unit: kilo] | 82.4 [54 to 101] | 62.8 [45 to 78] | 67.9 [54 to 77] | 69.6 [44 to 86] | 74 [52 to 103] | 67.7 [63 to 76] | 80.6 [57 to 97] | 66.6 [43 to 89] | 69.6 [58 to 81] | 71.1 [43 to 103]

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Identification of DLT defined as an adverse event occurring during the first treatment cycle, judged to be related to MEN1112 and meeting any of the following criteria:
  * Grade 3 non-haematological toxicity lasting more than 7 days
  * Grade ≥ 4 non-haematological toxicity.
Time Frame: over 3 weeks after the first dose
Population: For 'Single shot' administration: All patients receiving at least 1st & 2nd drug administration (dose 0.1 and 0.3 mg/kg) or completing first Cycle (doses ≥ 0.6 mg/kg) and safety FU ≥ 6 days post last dose or having experienced a DLT For 'Ramp up'': All patients receiving at least 80% of the scheduled drug administration during 1st Cycle and with a safety FU ≥ 6 days post last dose or having experienced a DLT
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 3 | 6 | 6 | 7 | 18 | 5 | 3 | 3 | 3
Participants | 0 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Identification of MTD defined as one dose level below the Maximum Administered Dose (i.e. one dose level below the one at which ≥ 2 DLTs out of 6 treated patients occur).
Time Frame: over 3 weeks after the first dose
Population: All subjects who received at last one dose of study treatment
Measure: Number; unit: mg/kg
Groups:
- MEN1112: MEN1112 given as "one shot" infusion or "ramp up"
Arm/Group | MEN1112
Number analyzed (Participants) | 71
mg/kg | 1.7

3. Secondary Outcome: Treatment Emergent Signs and Symptoms (TESSs)
Description: Number of patients with Treatment Emergent Signs and Symptoms (TESSs) by CTCAE severity grade >3 and treatment related causality
Time Frame: 6 months
Population: All patients who received at least one dose of study treatment by dose cohort
Measure: Number; unit: participants
Groups:
- Cohort 1 (0.1 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 0.1 mg/kg
- Cohort 2 (0.3 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 0.3 mg/kg
- Cohort 2b (0.6 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 0.6 mg/kg
- Cohort 3 (1.0 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 1.0 mg/kg
- Cohort 3b (1.7 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 1.7 mg/kg
- Cohort 3c (2.5 mg/kg): MEN1112 given as "one shot" infusion at the dosage of 2.5 mg/kg
- Cohort 1.7 Ramp up: MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg
- Cohort 2.0 Ramp up: MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg
- Cohort 3.0 Ramp up: MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg
Arm/Group | Cohort 1 (0.1 mg/kg) | Cohort 2 (0.3 mg/kg) | Cohort 2b (0.6 mg/kg) | Cohort 3 (1.0 mg/kg) | Cohort 3b (1.7 mg/kg) | Cohort 3c (2.5 mg/kg) | Cohort 1.7 Ramp up | Cohort 2.0 Ramp up | Cohort 3.0 Ramp up
Number analyzed (Participants) | 4 | 7 | 6 | 8 | 26 | 5 | 3 | 8 | 4
participants
  Patients with TESSs of CTCAE severity grade > or =3 | 3 | 6 | 6 | 8 | 26 | 5 | 3 | 8 | 4
  Patients with treatment related TESSs of CTCAE severity grade > or =3 | 2 | 1 | 4 | 5 | 11 | 5 | 1 | 2 | 2

4. Secondary Outcome: MEN1112 Pharmacokinetic (PK) Parameter Cmax
Description: Cmax is the maximum serum drug concentration. For Cohort 1 to 3c (administration as 'one shot' infusion) Cmax is measured at the end of the first intravenous infusion ( 1 to 6 hours; depending on the individual subjects being the infusion frequently interrupted) For Cohort 1.7, 2.0 and 3.0 (dose administration as ramp up, divided in three sub-doses), Cmax is measured at the end of each out of 3 intravenous infusions
Time Frame: end of intravenous infusion
Population: patients with reliable PK blood samples available at the end of drug intravenous infusion for Cmax measurement
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Cohort 1.7 (0.1 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg - first dose (0.1 mg) of the 3 ramp up total dose
- Cohort 1.7 (0.6 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg - second dose (0.6 mg) of the 3 ramp up total dose
- Cohort 1.7 (1.0 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg - third dose (1.0 mg) of the 3 ramp up total dose
- Cohort 2.0 (0.1 mg Out of 2.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg- first dose (0.1 mg) of the 3 ramp total dose
- Cohort 2.0 (0.7 Out of 2.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg- second dose (0.7 mg) of the 3 ramp total dose
- Cohort 2 (1.2 Out of 2.0 mg): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg- third dose (1.2 mg) of the 3 ramp total dose
- Cohort 3.0 (0.2 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- first dose (0.2 mg) of the 3 ramp total dose
- Cohort 3.0 (1.0 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- second dose (1.0 mg) of the 3 ramp total dose
- Cohort 3.0 (1.8 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- third dose (1.8 mg) of the 3 ramp total dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 (0.1 Out of 1.7 mg/kg) | Cohort 1.7 (0.6 Out of 1.7 mg/kg) | Cohort 1.7 (1.0 Out of 1.7 mg/kg) | Cohort 2.0 (0.1 mg Out of 2.0 mg/kg) | Cohort 2.0 (0.7 Out of 2.0 mg/kg) | Cohort 2 (1.2 Out of 2.0 mg) | Cohort 3.0 (0.2 Out of 3.0 mg/kg) | Cohort 3.0 (1.0 Out of 3.0 mg/kg) | Cohort 3.0 (1.8 Out of 3.0 mg/kg)
Number analyzed (Participants) | 4 | 7 | 6 | 7 | 26 | 5 | 3 | 2 | 3 | 8 | 7 | 8 | 4 | 4 | 3
mcg/mL | 0.22 (0.32) | 1.86 (2.06) | 3.29 (1.87) | 9.29 (5.07) | 2.67 (15.73) | 31.59 (18.18) | 2.65 (4.49) | 11.8 (2.91) | 18.57 (8.54) | 0.97 (2.18) | 7.62 (1.59) | 17.53 (6.6) | 1.26 (0.96) | 14.83 (8.57) | 39.73 (20.44)

5. Secondary Outcome: MEN1112 PK Parameter AUC (0-t)
Description: AUC (0-t) is the area under the serum concentration-time curve from time 0 extrapolated to t time evaluated after the first dose
Time Frame: Dose 1- cycle 1
Population: population with reliable PK parameters
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Groups:
- Cohort 1.7 (0.1 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg- first dose (0.1 mg/kg) of 3 ramp up total dose
- Cohort 1.7 (0.6 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg- second dose (0.6 mg/kg) of 3 ramp up total dose
- Cohort 1.7 (1.0 Out of 1.7 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 1.7 mg/kg- third dose (1.0 mg/kg) out of 3 ramp up total dose
- Cohort 2.0 (0.1 Out of 2.0 mg): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg-- first dose (0.1 mg/kg) of 3 ramp up total dose
- Cohort 2.0 (0.7 Out of 2 mg/kg Ramp up): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg- second dose (0.7 mg/kg) of 3 ramp up total dose
- Cohort 2.0 (1.2 Out of 2.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 2.0 mg/kg- third dose (1.2 mg/kg) of 3 ramp up total dose
- Cohort 3.0 (0.2 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- first dose (0.2 mg/kg) of 3 ramp up total dose
- Cohort 3.0 (1.0 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- second dose (1.0 mg/kg) of 3 ramp up total dose
- Cohort 3.0 (1.8 Out of 3.0 mg/kg): MEN1112 given as "ramp-up" infusions at the dosage of 3.0 mg/kg- third dose (1.8 mg/kg) of 3 ramp up total dose
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 (0.1 Out of 1.7 mg/kg) | Cohort 1.7 (0.6 Out of 1.7 mg/kg) | Cohort 1.7 (1.0 Out of 1.7 mg/kg) | Cohort 2.0 (0.1 Out of 2.0 mg) | Cohort 2.0 (0.7 Out of 2 mg/kg Ramp up) | Cohort 2.0 (1.2 Out of 2.0 mg/kg) | Cohort 3.0 (0.2 Out of 3.0 mg/kg) | Cohort 3.0 (1.0 Out of 3.0 mg/kg) | Cohort 3.0 (1.8 Out of 3.0 mg/kg)
Number analyzed (Participants) | 2 | 6 | 6 | 7 | 26 | 5 | 2 | 2 | 3 | 7 | 7 | 8 | 4 | 4 | 3
h*mcg/mL | 0.47 (0.5) | 79.48 (80.69) | 74.11 (88.45) | 346.8 (288.82) | 891.09 (642.63) | 1791.32 (1525.94) | 62.53 (87.94) | 200.15 (79.17) | 940.48 (686.59) | 5.87 (10.55) | 115.1 (33.66) | 843.53 (518.65) | 18.67 (14.63) | 194.91 (103.12) | 2385.21 (1956.83)

6. Secondary Outcome: MEN1112 PK Parameter AUC (0-∞)
Description: AUC (0-∞) is the area under the serum concentration-time curve from time 0 extrapolated to infinite time
Time Frame: dose 1 of cycle 1
Population: all subjects with Pk concentrations allowing a reliable estimation of AUC (0-∞). NOTE: cohort 1 excluded because of non reliable estimation of AUC (0-∞)
Measure: Mean (Standard Error); unit: h*mcg/mL
Arm/Group | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 5 | 5 | 7 | 23 | 5 | 3 | 7 | 3
h*mcg/mL | 99.89 (81.08) | 90.55 (91.67) | 370.69 (318.5) | 1321.55 (800.89) | 2220.48 (2009.55) | 1310.79 (1091.61) | 1516.51 (867.13) | 3894.85 (3352.56)

7. Secondary Outcome: MEN1112 PK Parameter t1/2
Description: t1/2 is the drug elimination half-life
  It is calculated on the first dose for all cohorts
Time Frame: dose 1 of cycle 1
Population: PK population with drug measurment allowing reliable estimation of half-life (cohort 1 excluded since estimation of half-life as well as AUC 0-inf was not reliable)
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 5 | 5 | 7 | 23 | 5 | 3 | 7 | 3
hour | 18.63 (6.47) | 10.76 (9.22) | 21.21 (15.05) | 46.49 (34.25) | 38.34 (26.72) | 46.84 (35.2) | 72.51 (46.88) | 61.75 (30.75)

8. Secondary Outcome: Complete Remission (CR) Rate
Description: CR rate at any time point, where CR is defined as: bone marrow blasts <5%, absence of extramedullary disease, absolute neutrophil count >1 x 109/L and platelet count > 100 x 109/L.
  According to the protocol, the efficacy analysis population includes all patients completing the first treatment cycle and having a post-cycle peripheral blood lab test and bone marrow aspirate.
Time Frame: 6 months
Population: According to the protocol, the efficacy analysis population includes all patients completing the first treatment cycle and having a post-cycle peripheral blood lab test and bone marrow aspirate.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 2 | 4 | 5 | 5 | 15 | 3 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Best Response Rate
Description: best observed response at any time point to include Complete Remission (CR is defined as bone marrow blasts < 5%, absence of extramedullary disease, absolute neutrophil count > 1 x 109 / L and platelet count > 100 x 109 / L) Complete Remission with incomplete blood count recovery [CRi defined as all criteria for CR except residual thrombocytopenia (platelets <100 x 109/L), and/or neutropenia (absolute neutrophil count <1 x 109/L)] Partial remission (PR defined as all haematological criteria for CR with bone marrow blasts 5-25% and decrease of pre-treatment bone marrow blast percentage by at least 50%.
Time Frame: 6 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 2 | 4 | 5 | 5 | 15 | 3 | 1 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) is the time from the date of the first drug administration to the date of death from any cause. If the fatal event does not occur during the study, the overall survival time is censored at the date when the patient was last known to be alive.
  The overall survival (OS) is calculated on 29 patients (72.5%) out of 40 belonging to the efficacy population.
  Results are reported as mean (and range) days
Time Frame: 6 months
Population: Overall Survival (OS) is the time from the date of the first drug administration to the date of death from any cause. If the fatal event does not occur during the study, the overall survival time is censored at the date when the patient was last known to be alive.
  The overall survival (OS) is calculated on 29 patients (72.5%) out of 40 belonging to the efficacy population. OS(measured in days) is reported as mean (and range)
Measure: Mean (Full Range); unit: day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 2b | Cohort 3 | Cohort 3b | Cohort 3c | Cohort 1.7 | Cohort 2.0 | Cohort 3.0
Number analyzed (Participants) | 2 | 4 | 5 | 5 | 15 | 3 | 1 | 3 | 2
day | 33 [33 to 33] | 56.5 [46.0 to 67] | 76.8 [30 to 123] | 47 [33 to 73] | 55.2 [24 to 129] | 92 [76 to 108] | 30 [30 to 30] | 52.5 [29 to 76] | 37 [28 to 46]

11. Other Pre Specified Outcome: Immunogenicity of MEN1112
Description: Incidence of anti-MEN1112 auto-antibodies
Time Frame: 64 days
Population: Analysis of immunogenicity was not done in any patients participating to the study, since no clinical benefit was detected in any patients under the experimental conditions adopted in the study; the study was terminated
Groups:
- MEN1112: Incidence of immunogenicity to be evaluated at the end of the treatment administration (day 64) was part of the secondary end-point. Due to study termination, immunogenicity analysis was not performed
Arm/Group | MEN1112
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were to be collected for 180 days (i.e. from Informed Consent signature to the End of Study Visit) or 70 days after last study drug administration whichever occurs last.
Arm/Group | Cohort 1 (0.1 mg/kg) | Cohort 2 (0.3 mg/kg) | Cohort 2b (0.6 mg/kg) | Cohort 3 (1.0 mg/kg) | Cohort 3b (1.7 mg/kg) | Cohort 3c (2.5 mg/kg) | Cohort 1.7 Ramp up | Cohort 2.0 Ramp up | Cohort 3.0 Ramp up
All-Cause Mortality (participants affected / at risk) | 3/4 | 4/7 | 5/6 | 8/8 | 17/26 | 4/5 | 2/3 | 5/8 | 3/4
Serious Adverse Events (participants affected / at risk) | 3/4 | 5/7 | 6/6 | 8/8 | 25/26 | 5/5 | 2/3 | 8/8 | 4/4
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 6/6 | 8/8 | 26/26 | 5/5 | 3/3 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.1 mg/kg) (N=4) | Cohort 2 (0.3 mg/kg) (N=7) | Cohort 2b (0.6 mg/kg) (N=6) | Cohort 3 (1.0 mg/kg) (N=8) | Cohort 3b (1.7 mg/kg) (N=26) | Cohort 3c (2.5 mg/kg) (N=5) | Cohort 1.7 Ramp up (N=3) | Cohort 2.0 Ramp up (N=8) | Cohort 3.0 Ramp up (N=4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 3 | 14 | 1 | 1 | 2 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 2 | 1 | 0 | 5 | 1 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anorectal cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 2 | 1 | 0 | 2 | 4 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.1 mg/kg) (N=4) | Cohort 2 (0.3 mg/kg) (N=7) | Cohort 2b (0.6 mg/kg) (N=6) | Cohort 3 (1.0 mg/kg) (N=8) | Cohort 3b (1.7 mg/kg) (N=26) | Cohort 3c (2.5 mg/kg) (N=5) | Cohort 1.7 Ramp up (N=3) | Cohort 2.0 Ramp up (N=8) | Cohort 3.0 Ramp up (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 4 | 2 | 11 | 0 | 2 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2 | 4 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 6 | 0 | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 9 | 0 | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intraocular haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 5 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 6 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 6 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 4 | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 8 | 0 | 0 | 1 | 0
Catheter site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 1 | 4 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 4 | 1 | 4 | 3 | 0 | 1 | 2 | 2
Biliary dilatation (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Graft versus host disease in liver (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemodilution (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 2 | 15 | 3 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 3 | 3 | 1 | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2 | 5 | 0 | 1 | 3 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Interleukin level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1
Procalcitonin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 4 | 2 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2 | 8 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 6 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 5 | 0 | 2 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 5 | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Central-alveolar hypoventilation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 3 | 2 | 0 | 5 | 1 | 1 | 0 | 2
Neurological symptom (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study terminated due to any clinical objective response observed in the patients' study population and under the study procedures implemented in the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the Investigator will allow Menarini Ricerche S.p.A. at least 30-day time to review and comment upon the publication manuscript. Menarini Ricerche S.p.A.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT02353143/Prot_SAP_000.pdf